CLINICAL TRIAL: NCT06883578
Title: Effect of Low Valine Diet on Body Weight and Metabolic Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2024-402R
Record Dates: First submitted 2025-03-09; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Overweight/obesity; Metabolic Associated Fatty Liver Disease; Metabolic Diseases
Keywords: Obesity; Dietary intervention; Low valine meal replacement
MeSH Terms: conditions — Overweight; Obesity; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Eligible subjects were enrolled according to the inclusion criteria. They will be enrolled into short-term continuous intervention or long-term intermittent intervention program according to their wishes, until the subjects of the intervention program are full.The subjects of the short-term 2-week continuous intervention or long-term 16-week intermittent intervention studies will be randomly assigned into the control meal replacement group and the low valine meal replacement group by random allocation separately, with 12 people in each group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Short-term continuous normal meal replacement intervention group (Placebo Comparator): The normal meal replacement intake is calculated at 25kcal/kg body weight per person per day, with the calorie ratio for breakfast, lunch and dinner being 1:2:2. A meal replacement diet is given for 2 consecutive weeks.
  Interventions: Dietary Supplement: Short-term continuous normal meal replacement
- Short-term continuous low valine meal replacement intervention group (Experimental): The low valine meal replacement intake is calculated at 25kcal/kg body weight per person per day, with the calorie ratio for breakfast, lunch and dinner being 1:2:2. A meal replacement diet is given for 2 consecutive weeks.
  Interventions: Dietary Supplement: Short-term continuous low-valine meal replacements
- Long-term intermittent normal meal replacement intervention group (Placebo Comparator): The normal meal replacement intake was calculated at 25 kcal/kg body weight per person per day, with the calorie distribution ratio of 1:2:2 for breakfast, lunch and dinner. A meal replacement diet was used for 2 consecutive days per week for 16 consecutive weeks.
  Interventions: Dietary Supplement: Long-term intermittent normal meal replacement
- Long-term intermittent low valine meal replacement intervention group (Experimental): The low valine meal replacement intake was calculated at 25 kcal/kg body weight per person per day, with the calorie distribution ratio of 1:2:2 for breakfast, lunch and dinner. A meal replacement diet was used for 2 consecutive days per week for 16 consecutive weeks.
  Interventions: Dietary Supplement: Long-term intermittent low valine meal replacement

INTERVENTIONS:
Dietary Supplement: Short-term continuous normal meal replacement — The normal meal replacement intake is calculated at 25kcal/kg body weight per person per day, with the calorie ratio for breakfast, lunch and dinner being 1:2:2. A meal replacement diet is given for 2 consecutive weeks.
  Arms: Short-term continuous normal meal replacement intervention group
Dietary Supplement: Short-term continuous low-valine meal replacements — The low valine meal replacement intake is calculated at 25kcal/kg body weight per person per day, with the calorie ratio for breakfast, lunch and dinner being 1:2:2. A meal replacement diet is given for 2 consecutive weeks.
  Arms: Short-term continuous low valine meal replacement intervention group
Dietary Supplement: Long-term intermittent normal meal replacement — The normal meal replacement intake was calculated at 25 kcal/kg body weight per person per day, with the calorie distribution ratio of 1:2:2 for breakfast, lunch and dinner. A meal replacement diet was used for 2 consecutive days per week for 16 consecutive weeks.
  Arms: Long-term intermittent normal meal replacement intervention group
Dietary Supplement: Long-term intermittent low valine meal replacement — The low valine meal replacement intake was calculated at 25 kcal/kg body weight per person per day, with the calorie distribution ratio of 1:2:2 for breakfast, lunch and dinner. A meal replacement diet was used for 2 consecutive days per week for 16 consecutive weeks.
  Arms: Long-term intermittent low valine meal replacement intervention group

SUMMARY:
This study aimed to explore the effects of ordinary meal replacements and low-valine meal replacements on the weight and risk of related metabolic diseases in overweight/obese patients through a randomized double-blind controlled clinical trial.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled clinical study, which aims to explore the advantages of low valine meal replacements in weight loss and improving metabolism compared with ordinary meal replacements. It is divided into two parts: 1) short-term continuous low valine meal replacement intervention (2 weeks) and 2) long-term intermittent low valine meal replacement intervention (16 weeks). Overweight and obese subjects will be enrolled according to the inclusion and exclusion criteria, and entered the short-term continuous intervention and long-term intermittent intervention projects according to the subjects' wishes until the number of subjects planned for the project is filled. The subjects of the short-term 2-week continuous intervention and long-term 16-week intermittent intervention studies will be randomly assigned to the control meal replacement group and the low valine meal replacement group by random allocation, with 12 people in each group.

The randomization sequence of this study will be generated by an independent statistician team based on the clinical research plan and random allocation parameter configuration file. During the generation process, all necessary information and related parameters, including system software version, random number seed, sequence length, block length, group information, inter-group ratio, stratification factors and levels, will be recorded in detail in the randomization table to ensure the reproducibility and reliability of randomization. All subjects and investigators (including members of the research team and the intervention implementers) are blind to the grouping of subjects during the study period.

The primary outcome is the change of body weight, which will be measured at baseline and at the end of follow-up. Secondary endpoints include changes in plasma glucose, serum lipid profiles, liver enzymes, and DXA body composition. For patients with long-term low-valine meal replacement intervention, liver fat content measured by PDFF will also be measured. At the same time, serum proteomic, metabolomic and lipidomic profiles of all subjects at the end of follow-up will be analyzed to preliminarily expand the study of the possible mechanism of low valine diet in regulating body weight.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 16 years old ≤ age ≤ 80 years old;
* BMI ≥ 24kg/m2

Exclusion Criteria:

* Excessive drinkers (defined as: in the past 6 months, the weekly alcohol intake of men exceeds 140g, and that of women exceeds 70g);
* Liver diseases caused by other reasons: such as alcoholic liver disease, acute and chronic viral hepatitis, drug-induced, immune hepatitis (AMA, SMA, ANA), cirrhosis, liver cancer, etc.;
* Other diseases that affect glucose and lipid metabolism: hyperthyroidism, hypothyroidism, Cushing's syndrome, etc.;
* Poorly controlled diabetic patients: HbA1c >9.5% within three months; or use of hypoglycemic drugs that may affect weight, including pioglitazone, GLP-1, SGLT2 inhibitors;
* Chronic kidney disease or severe renal impairment, defined as serum creatinine greater than 2.0mg/dL;
* Serum ALT greater than 3 times the upper limit of normal;
* Life expectancy of no more than 3 years in the presence of serious health conditions;
* Those who plan to get pregnant in the near future;
* Those who cannot participate in the follow-up of the intervention due to other conditions;
* Continuously used drugs that may cause weight changes for more than 2 weeks in the past year (such as glucocorticoids, thyroid hormones, etc.);
* Participated in other clinical trials in the past 4 weeks;
* Those who had gastric volume reduction surgery or digestive tract surgery;
* Those diagnosed with any tumor disease;
* Subjects who participated in strenuous exercise or planned to change their diet structure;
* Unable to sign the informed consent form.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | From enrollment to the end of intervention at 2 weeks or 16 weeks

SECONDARY OUTCOMES:
Fat mass | From enrollment to the end of intervention at 2 weeks or 16 weeks
Lean mass | From enrollment to the end of intervention at 2 weeks or 16 weeks
Fasting plasma glucose | From enrollment to the end of intervention at 2 weeks or 16 weeks
2h postload plasma glucose | From enrollment to the end of intervention at 2 weeks or 16 weeks
Fasting insulin | From enrollment to the end of intervention at 2 weeks or 16 weeks
2h postload insulin | From enrollment to the end of intervention at 2 weeks or 16 weeks
Triglycerides | From enrollment to the end of intervention at 2 weeks or 16 weeks
Cholesterol | From enrollment to the end of intervention at 2 weeks or 16 weeks
LDL cholesterol | From enrollment to the end of intervention at 2 weeks or 16 weeks
HDL cholesterol | From enrollment to the end of intervention at 2 weeks or 16 weeks
Total bilirubin | From enrollment to the end of intervention at 2 weeks or 16 weeks
Conjugated bilirubin | From enrollment to the end of intervention at 2 weeks or 16 weeks
Creatinine | From enrollment to the end of intervention at 2 weeks or 16 weeks
Uric acid | From enrollment to the end of intervention at 2 weeks or 16 weeks
Systolic blood pressure | From enrollment to the end of intervention at 2 weeks or 16 weeks
Diastolic blood pressure | From enrollment to the end of intervention at 2 weeks or 16 weeks
Waist circumference | From enrollment to the end of intervention at 2 weeks or 16 weeks
HbA1c | From enrollment to the end of intervention at 2 weeks or 16 weeks
  Measured only in long-term intermittent intervention subjects
PDFF liver fat content | From enrollment to the end of intervention at 16 weeks
  Measured only in long-term intermittent intervention subjects

OTHER OUTCOMES:
Serum proteomic profiles | From enrollment to the end of intervention at 2 weeks or 16 weeks
Serum metabolomic profiles | From enrollment to the end of intervention at 2 weeks or 16 weeks
Serum lipidomic profiles | From enrollment to the end of intervention at 2 weeks or 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/